CLINICAL TRIAL: NCT05893537
Title: A Randomized, Double-Masked, Placebo-Controlled, Parallel-Group, Phase 2 Study to Evaluate the Efficacy and Safety of Oral CT1812 in Participants With Geographic Atrophy (GA) Secondary to Dry Age-Related Macular Degeneration (AMD).
Brief Title: Study to Evaluate the Efficacy and Safety of Oral CT1812 in Participants With Geographic Atrophy (GA) Secondary to Dry Age-Related Macular Degeneration (AMD).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was closed as part of a strategic business decision.
Sponsor: Cognition Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG2201
Record Dates: First submitted 2023-05-17; First posted 2023-06-08 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-03

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT1812 200 mg (Active Comparator): Drug: CT1812 Active Study Drug
  Interventions: Drug: Active Comparator CT1812
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Active Comparator CT1812 — 123 participants will receive a single daily dose of CT1812 (200 mg)
  Arms: CT1812 200 mg
Drug: Placebo Comparator — 123 participants will receive a single daily dose of placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, prospective, multicenter, randomized, double-masked, placebo-controlled 104-week study to assess the efficacy, safety, and tolerability of orally delivered CT1812 compared to placebo in participants with GA associated with dry AMD.

DETAILED DESCRIPTION:
This is a Phase 2, prospective, multicenter, randomized, double-masked, placebo-controlled 104-week study to assess the efficacy, safety, and tolerability of orally delivered CT1812 compared to placebo in participants with GA associated with dry AMD.

Participants ≥50 years old diagnosed with GA secondary to dry AMD and who meet all inclusion criteria and none of the exclusion criteria will be included in the study. The study will randomize up to 246 participants in a 1:1 manner (123 participants per treatment group) to receive a single daily dose of either CT1812 (200 mg) or placebo across approximately 40-50 sites.

Following a screening period of up to 60 days, the total expected duration of participant participation in the study will be 108 weeks (104-week treatment period followed by a 28-day [4-week] post treatment safety follow up period).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years at time of informed consent.
2. BCVA of 24 letters or better using Early Treatment Diabetic Retinopathy Study (ETDRS) charts at screening.
3. Stable pharmacological treatment of any other chronic conditions for at least 30 days prior to screening.

EXCLUSION CRITERIA:

1. GA due to causes other than dry AMD.
2. Any history or current evidence of exudative ("wet") AMD.
3. Retinal disease other than dry AMD.
4. Any ophthalmologic condition that prevents adequate imaging of the retina as judged by the study site or central reading center.
5. Intraocular surgery (including intraocular lens implantation surgery) within 3 months prior to randomization.
6. Any ophthalmic condition that will or is likely to require surgery during the study period.
7. Hypersensitivity to fluorescein.
8. Suspected or known allergy to any components of the study treatments.
9. History of vitrectomy surgery, submacular surgery or any other surgical intervention for dry AMD.
10. History of glaucoma filtering surgery or corneal transplant in the study eye.
11. History of central serous retinopathy in either eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Geographic Atrophy (GA) lesion area over 104 weeks in the study eye. | Baseline through Week 104
  Compare the mean rate of growth (slope) in GA lesion area in the study eye measured by fundus autofluorescence imaging (FAF).

SECONDARY OUTCOMES:
Safety and Tolerability of CT1812 | Baseline through Week 104
  Incidence and Severity of Adverse Events compared to placebo in participants with GA secondary to dry AMD.
Plasma concentration of CT1812 | Baseline through Week 104
  Measure pre-dose plasma concentration of CT1812.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, Study Director — Cognition Therapeutics Inc.
Locations (19):
- United States (19):
  - Phoenix Retina Associates, Phoenix, Arizona
  - Retinal Consultants Medical Group, Sacramento, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Advanced Research, Deerfield Beach, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Retina Specialists, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - NJ Retina, Edison, New Jersey
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Verum Research LLC, Eugene, Oregon
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Tennessee Retina, PC, Nashville, Tennessee
  - Austin Clinical Research, LLC, Austin, Texas
  - Star Vision Consultants, Burleson, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Retina Consultants of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Magnify Study — http://magnifydryamdstudy.com